CLINICAL TRIAL: NCT03009227
Title: Study of Oncological Outcomes of D3 Lymph Node Dissection in Colon Cancer
Acronym: COLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: N.N. Petrov National Medical Research Center of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COL-1
Record Dates: First submitted 2016-12-29; First posted 2017-01-04 (Estimated); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Colonic Neoplasms Malignant
Keywords: colon cancer; lymph node dissection; D3 lymph node dissection
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D2 lymph node dissection (Active Comparator): Colonic resection with D2 lymph node dissection
  Interventions: Procedure: Colonic resection with D2 lymph node dissection
- D3 lymph node dissection (Experimental): Colonic resection with D3 lymph node dissection
  Interventions: Procedure: Colonic resection with D3 lymph node dissection

INTERVENTIONS:
Procedure: Colonic resection with D2 lymph node dissection — Appropriate to the tumor location colonic resection is performed with D2 lymph node dissection
  Arms: D2 lymph node dissection
Procedure: Colonic resection with D3 lymph node dissection — Appropriate to the tumor location colonic resection is performed with D3 lymph node dissection
  Arms: D3 lymph node dissection

SUMMARY:
The purpose of this study is to determine wether D3 lymph node dissection gives superior oncological outcomes compared to standard D2 lymph node dissection in colon cancer

DETAILED DESCRIPTION:
The design involves random allocation of eligible patients to D3 or D2 lymph node dissection group in 1:1 ratio. The extent of colonic resection itself is not influenced by the randomization and is predefined by the investigator prior to randomization.

Requirements applied to centers participating in the trial and surgeons performing procedures are described in the protocol and refer to center volume and surgeon's experience with evaluation of non-edited video-recordings of procedures.

Routine quality control includes requirement to photograph vessels with the clip to determine the extent of lymph node dissection performed and a thorough morphological assessment of the specimen.

After surgery patients are treated according to local standards with no difference wether D2 or D3 lymph node dissection was performed. Short-term and long-term outcomes are registered as per protocol.

This is a superiority trial evaluating statistical superiority. With the 50% five year survival according to national registry for colon cancer, expecting 10% improvement in survival with D3 lymph node dissection, enrollment of 768 patients during 3 year accrual period followed by 5 year follow up is required for a power of 80%.

The intent-to-treat principle is used for the data analysis.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed adenocarcinoma of the colon (caecum, ascending, transverse, descending, sigmoid)
* clinical stage T1-4aN0-2M0-1 (distant metastases must be resectable)
* indications for surgical colonic resection
* ECOG status 0-2
* At least 18 years of age
* Written informed consent

Exclusion Criteria:

* Medical or psychiatric conditions that compromise the patient's ability to give informed consent or comply with the study protocol
* Pregnancy or breast feeding
* Medical contraindications for surgical treatment
* Synchronous or metachronous malignancy
* Non-resectable distant metastases
* Colon obstruction, perforation or bleeding complicating the tumor
* Indications for isolated transverse colon resection
* Neoadjuvant chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years after last patient enrolled
  overall survival of patients

SECONDARY OUTCOMES:
Disease-free survival | 5 years after last patient enrolled
  Survival without local or systemic recurrence
Postoperative morbidity | within the first 30 days after surgery
  Complications after surgery
Postoperative mortality | within the first 30 days after surgery
  Death after surgery
Postoperative recovery parameters | within the first 30 days after surgery
  Complex of parameters describing the pattern of recovery after surgery (i.e. food tolerance, peristalsis, walking etc.)
Pattern of lymph node metastasis based on pathology report | enrollment period
  Number of lymph node with metastases related to number of lymph nodes studied in each group in the specimen
CME quality | enrollment period
  Ratio of good, satisfactory and unsatisfactory quality according to pathology report
Lymph node yield | enrollment period
  Number of lymph nodes removed according to pathology report
Quality of life in patients after D2 and D3 lymph node dissection using questionnaire | enrollment period
  CR29 and CR30 questionnaires by European Organization for Research and Treatment of Cancer

CONTACTS AND LOCATIONS:
Overall Officials: Aleksei Karachun, Ph.D., Study Chair — N.N. Petrov Research Institute of Oncology, Surgical department of abdominal oncology, St. Petersburg, Russian Federation
Locations (12):
- Russia (12):
  - Krasnodar City clinical hospital #1, Krasnodar
  - State Scientific Centre of Coloproctology, Moscow
  - Moscow city oncological hospital #62, Moscow
  - P. Herzen Moscow Oncology Research Institute, Moscow
  - Medical radiological scientific center named after A.F. Tsyba, Obninsk
  - Rostov Research Institute of Oncology, Rostov
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - St Petersburg City Clinical Oncology Dispensary, Saint Petersburg
  - Saint-Petersburg Clinical Research center of specialized kinds of medical care (Oncology), Saint Petersburg
  - Scientific-Research institute of Oncology named after N.N. Petrov, Saint Petersburg
  - Saint-Petersburg State University Clinic, Saint Petersburg
  - Republican clinical oncological dispencery, Ufa

IPD SHARING:
Plan to Share IPD: No
We are not planning to share personal patient data

REFERENCES:
- [Background] Karachun A, Petrov A, Panaiotti L, Voschinin Y, Ovchinnikova T. Protocol for a multicentre randomized clinical trial comparing oncological outcomes of D2 versus D3 lymph node dissection in colonic cancer (COLD trial). BJS Open. 2019 Mar 14;3(3):288-298. doi: 10.1002/bjs5.50142. eCollection 2019 Jun. PMID 31183444
- [Result] Karachun A, Panaiotti L, Chernikovskiy I, Achkasov S, Gevorkyan Y, Savanovich N, Sharygin G, Markushin L, Sushkov O, Aleshin D, Shakhmatov D, Nazarov I, Muratov I, Maynovskaya O, Olkina A, Lankov T, Ovchinnikova T, Kharagezov D, Kaymakchi D, Milakin A, Petrov A. Short-term outcomes of a multicentre randomized clinical trial comparing D2 versus D3 lymph node dissection for colonic cancer (COLD trial). Br J Surg. 2020 Apr;107(5):499-508. doi: 10.1002/bjs.11387. Epub 2019 Dec 24. PMID 31872869